CLINICAL TRIAL: NCT01083576
Title: Double-blind, Randomized, Pharmacokinetics, Safety, and Efficacy Trial of WR 279,396 (Paromomycin + Gentamicin Topical Cream) and Paromomycin Topical Cream for the Treatment of Cutaneous Leishmaniasis in Panama
Brief Title: Pharmacokinetics, Safety, and Efficacy Trial of WR 279,396 (Paromomycin + Gentamicin Topical Cream) and Paromomycin Topical Cream for the Treatment of Cutaneous Leishmaniasis in Panama
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PG-PANAMA-08-04; A-15810
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2014-05

CONDITIONS: Leishmaniasis, Cutaneous
Keywords: leishmaniasis; cutaneous; WR 279,396; paromomycin; gentamicin; pharmacokinetics; safety; efficacy
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis | interventions — Paromomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paromomycin Alone Treatment (Active Comparator): Paromomycin Alone Cream (15% paromomycin topical cream): topical application to uncomplicated cutaneous leishmaniasis (CL) lesions once daily for 20 days
  Interventions: Drug: Paromomycin Alone Cream (15% paromomycin topical cream)
- WR 279,396 (Active Comparator): WR 279,396 (15% paromomycin + 0.5% gentamicin topical cream): topical application to uncomplicated CL lesions once daily for 20 days
  Interventions: Drug: WR 279,396 (15% paromomycin + 0.5% gentamicin topical cream)

INTERVENTIONS:
Drug: WR 279,396 (15% paromomycin + 0.5% gentamicin topical cream) — topical application to CL lesions once daily for 20 days
  Other Names: Topical paromomycin/gentimicin cream
  Arms: WR 279,396
Drug: Paromomycin Alone Cream (15% paromomycin topical cream) — topical application to CL lesions once daily for 20 days
  Arms: Paromomycin Alone Treatment

SUMMARY:
The objectives of the study are to evaluate the pharmacokinetics (PK), safety, and efficacy of WR 279,396 (Paromomycin + Gentamicin Topical Cream) and Paromomycin Topical Cream in subjects with cutaneous leishmaniasis (CL).

DETAILED DESCRIPTION:
This study is a single-site, randomized, double-blind, two group trial assessing the PK, safety and efficacy of WR 279,396 Topical Cream and Paromomycin Topical Cream in subjects with CL. Subjects will be screened over a period up to 28 days for eligibility including parasitology for confirmation of ulcerative CL. Subjects will be randomized in a targeted 1:1 ratio to receive either WR 279,396 (15% paromomycin + 0.5% gentamicin topical cream) (target n=15) or Paromomycin Topical Cream (15% paromomycin topical cream) (target n=15) by topical application to CL lesions once daily for 20 days. Because the primary objective of this trial is to determine PK in all age groups, subjects will be stratified by age: 5-11 yrs, 12-17 yrs, and ≥ 18 yrs with at least 6 PK subjects in each age stratum and no more than 18 total subjects will be randomized in any age range. A target of 30 subjects who complete the PK part of the study is the goal. Any subject who does not complete the PK portion of the study will be replaced with another subject from the same age group that will be given the same treatment assignment to maintain the balance. Safety will be assessed by monitoring adverse events (AEs), lesion site reactions, vital signs, and blood creatinine levels. The primary efficacy analysis will be by evaluation of an index lesion with secondary efficacy analyses including all lesions. Lesions will also be examined for parasite negativity by classical means (positive culture for promastigotes or microscopic identification of amastigotes in stained lesion tissue) on Day 21.

In adult subjects, on Days 1 and 20, blood will be collected prior to topical cream application and at 0.5h, 1h, 2h, 3h, and 4h ± 5 minutes and 8h, 12h, and 24h ± 15 minutes after completion of cream application to determine plasma levels of paromomycin and gentamicin to calculate PK parameters. Thus, the last blood draw in this series will occur on Day 21. In addition, blood will be collected on Days 4, 7, 12, and 17 ± 1 day before study drug application to examine trough plasma levels of paromomycin and gentamicin. A follow-up plasma sample for PK analysis will also be obtained on Day 28 ± 2 days.

Subjects under the age of 18 years will have a total of four blood samples drawn. The first will be drawn at pre-application and the second will be drawn at 4 hours ± 5 minutes after completion of application of the topical cream on Study Day 1. The third will be drawn pre-application and the fourth at 4 hours ± 5 minutes after completion of application of the topical cream on Study Day 20. Subjects who receive Paromomycin Topical Cream are not expected to have blood levels of gentamicin, but as the study is blinded, plasma specimens will be tested for both paromomycin and gentamicin.

The index lesion (primary ulcerated) and all other ulcerated lesions will be assessed for clinical response by measurement of the length and width of area of ulceration. A lesion will be considered to be completely cured if 100% re-epithelialization is observed (i.e., this is a measurement of ulceration of 0 x 0 mm). Non-ulcerated lesions will also be measured to monitor the total area of exposure of lesions to study drug and will be evaluated for cure (i.e., absence of signs of an active lesion).

Subjects will have an in-clinic follow-up weekly (Days 28, 35, 42, 49, 56, and 63 ± 2 days) after completion of treatment for safety assessments, lesion measurements, and lesion photographs. On Day 21, index lesions in adult subjects that have not completely re-epithelialized will be assessed for parasites by classical means (positive culture for promastigotes or microscopic identification of amastigotes in stained lesion tissue). An interim analysis of all of the data collected on all subjects who were randomized and completed the nominal Day 63 follow-up will be performed to make decisions about the final design of a Phase 3 trial. Subjects will continue to be followed for outcomes at Day 100 and 168 ± 14 days. A final analysis of outcomes after the longer term followup period has been completed for all subjects will be performed when the trial is closed. Follow-up evaluations include AEs, medication use, lesion measurements, and lesion photographs.

Patients who fail therapy (see definition of failure below) may be administered rescue therapy at the discretion of the patient's personal physician.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, the following must be answered "YES" or not applicable, as appropriate for the study subject:

  1. Is the subject a male or female at least 5 years-of-age?
  2. Is the subject or legal guardian able to give written informed consent or assent, as appropriate?
  3. Does the subject have a diagnosis of CL in at least one lesion by at least one of the following methods: 1) positive culture for promastigotes, or 2) microscopic identification of amastigotes in stained lesion tissue.
  4. Does the subject have at least one ulcerative lesion ≥ 1 cm and ≤ 5 cm, that meets the criteria for an index lesion?
  5. Is the subject willing to forego other forms of treatments for CL including other investigational treatments during the study?
  6. In the opinion of the investigator, is the subject (or their legal guardian) capable of understanding and complying with the protocol?
  7. If female and of child-bearing potential, did the subject have a negative pregnancy test during screening and agree to use an acceptable method of birth control during the treatment phase and for 1 month after treatment is completed?
  8. Does the subject have adequate venous access for blood draws?

Exclusion Criteria:

To be eligible for the study, the following must be answered "NO" or not applicable as appropriate for the study subject:

1. Does the subject have only a single lesion whose characteristics include any of the following: verrucous or nodular lesion (non-ulcerative), lesion <1 cm in its greatest diameter, lesion in a location that in the opinion of the Investigator is difficult to maintain application of study drugs topically?
2. Does the subject have a lesion due to leishmania that involves the mucosa or palate or any signs of mucosal disease that might be due to leishmania?
3. Does the subject have signs and symptoms of disseminated disease in the opinion of the Principal Investigator?
4. Does the subject have > 10 lesions?
5. Is the subject a female who is breast-feeding?
6. Does the subject have an active malignancy or history of solid, metastatic or hematologic malignancy with the exception of basal or squamous cell carcinoma of the skin that has been removed?
7. Does the subject have significant organ abnormality, chronic disease such as diabetes, severe hearing loss, evidence of renal or hepatic dysfunction, or creatinine, aspartate aminotransferase (AST), or alanine aminotransferase (ALT) greater than 15% above the upper limit of normal (ULN) as defined by the clinical laboratory defined normal ranges?
8. Has the subject received treatment for leishmaniasis including any medication with pentavalent antimony including sodium stibogluconate (Pentostam), meglumine antimoniate (Glucantime); amphotericin B (including liposomal amphotericin B and amphotericin B deoxycholate); or other medications containing paromomycin (administered parenterally or topically) or methylbenzethonium chloride (MBCL); gentamicin; fluconazole; ketoconazole; pentamidine; miltefosine, azithromycin or allopurinol that was completed within 8 weeks of starting study treatments?
9. Does the subject have a history of known or suspected hypersensitivity or idiosyncratic reactions to aminoglycosides?
10. Does the subject have any other topical disease/condition which would interfere with the objectives of this study?

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Sosa, M.D. FACP, Principal Investigator — Instituto Conmemorativo Gorgas de Estudios de la Salud
Locations (1):
- Gorgas Memorial Institute Clinical Research Unit, Panama City, Panama

REFERENCES:
- [Derived] Ravis WR, Llanos-Cuentas A, Sosa N, Kreishman-Deitrick M, Kopydlowski KM, Nielsen C, Smith KS, Smith PL, Ransom JH, Lin YJ, Grogl M. Pharmacokinetics and absorption of paromomycin and gentamicin from topical creams used to treat cutaneous leishmaniasis. Antimicrob Agents Chemother. 2013 Oct;57(10):4809-15. doi: 10.1128/AAC.00628-13. Epub 2013 Jul 22. PMID 23877689

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Started | 15 | 15
Completed | 9 | 14
Not Completed | 6 | 1
Not completed — Treatment Failure | 6 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects were included in the mITT Analysis. All subjects met criteria for the evaluable subset.
Groups:
- Paromomycin Alone Treatment: Paromomycin Alone Cream (15% paromomycin topical cream): topical application to uncomplicated CL lesions once daily for 20 days
- Total: Total of all reporting groups
Arm/Group | Paromomycin Alone Treatment | WR 279,396 | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (16.2) | 25.5 (15.9) | 24.7 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 13 | 11 | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  Mestizo | 14 (100) | 15 (93.3) | 29
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Obtained Final Clinical Cure of Index Lesion
Description: Number of participants who had initial clinical cure (100% re-epithelialization of index lesion by Day 63) OR initial clinical improvements (> 50% re-epithelialization of index lesion followed by Day 63 by 100% re-epithelialization of the index lesion on or before Day 100), AND no relapse of index lesion.
Time Frame: 168 days
Population: All randomized subjects were included in the mITT Analysis. All subjects met criteria for the evaluable subset.
Measure: Number; unit: Participants
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 15 | 15
Participants | 9 | 13

2. Secondary Outcome: Number of Participants Who Obtained a Modified Final Clinical Cure of All Lesions
Description: Final cure as defined by the primary outcome measure AND and cure of all other lesions by Day 168. (100% re-epithelialization of all ulcerated lesions and resolution of all other type of lesions)
Time Frame: 168 days
Population: All randomized subjects were included in the mITT Analysis. All subjects met criteria for the evaluable subset.
Measure: Number; unit: Participants
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 15 | 15
Participants | 8 | 13

3. Secondary Outcome: Detectable Paromomycin or Gentamicin Plasma Levels
Description: Proportion of subjects with any detectable Paromomycin or Gentamicin plasma levels on a study day when blood for PK was collected
Time Frame: 20 days
Population: Adults ages >= 17 years
Measure: Number; unit: Participants
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 8 | 9
Participants
  Any detectable gentamicin | 0 | 1
  Any detectable paromomycin | 8 | 8

4. Secondary Outcome: Paromomycin Plasma Concentrations in Adults
Description: Paromomycin plasma concentrations following administration of paromomycin alone or WR 279,396 in adults
Time Frame: Day 4 to Day 28
Population: Adults ages >= 17 years
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 8 | 9
ng/mL
  Day 4 | 0 (0) | 17.8 (38.0)
  Day 7 | 13.1 (37.1) | 17.6 (34.9)
  Day 12 | 6.6 (18.8) | 26.4 (40.8)
  Day 17 | 44.0 (49.8) | 26.3 (52.3)
  Day 20 | 54.6 (48.4) | 31.4 (47.8)
  Day 28 | 0 (0) | 0 (0)

5. Secondary Outcome: Paromomycin Plasma Concentrations in Children
Description: Paromomycin plasma concentrations 4 hours following administration of paromomycin alone or WR 279,396 in children
Time Frame: Days 1 and 20
Population: Children ages 7 to 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 7 | 6
ng/mL
  Study Day 1 | 116.3 (83.6) | 98.6 (132.3)
  Study Day 20 | 992.7 (1149.7) | 634.2 (426.2)

6. Secondary Outcome: Pharmacokinetic Parameter: Cmax
Description: Cmax of paromomycin following administration of paromomycin alone or WR 279,396 to adults in Panama
Time Frame: 0, 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, 12.0, 24.0 hours on both Days 1 and 20
Population: Adults with measurable samples.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 8 | 9
ng/mL
  Day 1 | 219.0 (294) | 121 (106)
  Day 20 | 751.0 (609.0) | 561.0 (560.0)

7. Secondary Outcome: Pharmacokinetic Parameter: Tmax
Description: Tmax of paromomycin following administration of paromomycin alone or WR 279,396 to adults in Panama
Time Frame: 0, 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, 12.0, 24.0 hours on both Days 1 and 20
Population: Adults ages >= 17 years with measurable samples. Both groups had only 6 measureable samples each on Day 1.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 8 | 8
hr
  Day 1 | 2.7 (1.2) | 2.8 (2.6)
  Day 20 | 2.2 (0.8) | 2.2 (1.4)

8. Secondary Outcome: Pharmacokinetic Parameter: Area Under the Curve (AUC)
Description: Area under the curve (AUC) of paromomycin following administration of paromomycin alone or WR 279,396 to adults in Panama
Time Frame: 0, 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, 12.0, 24.0 hours on both Days 1 and 20
Population: Adults ages >= 17 years with measurable samples.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 8 | 9
ng*hr/mL
  Day 1 | 1571 (1850) | 863.4 (974.0)
  Day 20 | 5603 (4050) | 4740 (3987)

9. Other Pre Specified Outcome: Serum Creatinine Levels
Description: Blood creatinine was measured to assess possible nephrotoxicity associated with aminoglycosides
Time Frame: Day 1 and Day 20
Population: All randomized subjects were included in the mITT Analysis. All subjects met criteria for the evaluable subset.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 15 | 15
mg/dL
  Study Day 1 | 0.83 (0.23) | 0.79 (0.27)
  Study Day 20 | 0.77 (0.26) | 0.76 (0.22)

10. Secondary Outcome: Pharmacokinetic Parameter: t(1/2)
Description: t(1/2) of paromomycin following administration of paromomycin alone or WR 279,396 to adults in Panama
Time Frame: 0, 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, 12.0, 24.0 hours on both Days 1 and 20
Population: Adults ages >= 17 years with measurable samples. Paromomycin Alone Treatment had only 5 measureable samples on Day 1, and WR 279,396 had only 4 measureable samples on Day 20.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 7 | 8
hr
  Day 1 | 7.03 (7.67) | 4.0 (1.9)
  Day 20 | 5.3 (2.1) | 7.0 (3.6)

11. Secondary Outcome: Pharmacokinetic Parameter: Cmax/D
Description: Maximum observed plasma concentration divide by topical dose (Cmax/D) of paromomycin following administration of paromomycin alone or WR 279,396 to adults in Panama
Time Frame: 0, 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, 12.0, 24.0 hours on both Days 1 and 20
Population: Adults ages >= 17 years with measurable samples.
Measure: Mean (Standard Deviation); unit: 1/ML
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 8 | 9
1/ML
  Day 1 | 104.0 (104.0) | 61.3 (64.0)
  Day 20 | 227 (71) | 179 (128)

12. Secondary Outcome: Pharmacokinetic Parameter: AUC/D
Description: Area under the plasma concentration-time curve over 24 hrs divided by topical dose (AUC/D) of paromomycin following administration of paromomycin alone or WR 279,396 to adults in Panama
Time Frame: Days 1 and 20
Population: Adults ages >= 17 years with measurable samples.
Measure: Mean (Standard Deviation); unit: hr/ML
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 8 | 9
hr/ML
  Day 1 | 715.2 (748.1) | 345.9 (303.9)
  Day 20 | 1725 (530) | 1380 (631)

ADVERSE EVENTS:
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 14/15 | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paromomycin Alone Treatment (N=15) | WR 279,396 (N=15)
Application site erythema (General disorders) | 2 | 3
Application site oedema (General disorders) | 3 | 2
Application site pain (General disorders) | 5 | 1
Superinfection bacterial (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Mucocutaneous leishmaniasis (Infections and infestations) | 1 | 1
Burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 8 | 6

LIMITATIONS AND CAVEATS:
There are no PK tables for gentamicin due to low sample size; only 2 individuals with measureable gentamicin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No